CLINICAL TRIAL: NCT04661280
Title: Donepezil Use Versus Non-drug Approach in Treatment of Newly Diagnosed Alzheimer's Disease : a Multicentric, Randomized, Open Study : the CHOLINE-2 Study
Brief Title: Donepezil Versus Non-drug Treatment in Alzheimer's Disease.
Acronym: CHOLINE-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: France Alzheimer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP201183
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer Disease, Early Onset
Keywords: Alzheimer Disease; Donepezil
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive remediation (No Intervention): Non-drug treatment, cognitive remediation, cognitive stimulation
- Cognitive remediation + Donepezil (Experimental): Non-drug treatment, cognitive remediation, cognitive stimulation + Donepezil
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — Donepezil 5 mg per day during one month, then 10 mg per day during 5 months.
  Other Names: Aricept
  Arms: Cognitive remediation + Donepezil

SUMMARY:
Donepezil, as well as the other symptomatic drugs of Alzheimer's disease, is not any more reimbursed by the French healthcare system, due to a controversy about its efficiency. French health authorities currently preconize a non-rug approach based on cognitive remediation or stimulation.

The aim of this study is to compare the efficiency of the 2 approaches (non-drug versus donepezil) on the symptoms of Alzheimer's disease after 6 months of treatment.

DETAILED DESCRIPTION:
Randomized multicentric open-label study, comparison of 2 therapeutic strategies.

2 arms:

* Standard of care, non-drug approach: following the recommendations of the Alzheimer's disease care by the Frenchh Health Authority. The care is cognitive, psychic, functional or social and centered on the patient and his environment. This care is best carried out by the memory consultations participating in this study and having extensive experience in the care of Alzheimer patients. It is usually based in particular on the prescription of cognitive stimulation sessions by a speech therapist and a mobile Alzheimer specialist team at home for cognitive remediation sessions.
* Donepezil group: Management similar to the previous arm plus addition of Donepezil 5 mg per os once a day for one month and then 10 mg per os once a day until the 6th month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's disease according to the IWG-2 criteria.
* Age ≥ 50 years.
* Absence of legal protection measures (guardianship, curatorship).
* MMSE score ≥ 10 at inclusion.
* abnormal values for Aβ42 in the CSF or Aβ40 / Aβ42 ratio.
* abnormal values for phosphorylated Tau in CSF
* Presence of a family carer or a person at home who can ensure compliance with treatment if MMSE score <20.
* French native speaker.

Exclusion Criteria:

* Other cause of dementia.
* Previous use of symptomatic treatment for Alzheimer's disease.
* Hypersensitivity to donepezil hydrochloride or to any of the excipients listed in the SPC.
* Cardiological contraindication after possible opinion of a cardiologist, at the initiative of the investigator, in particular bradycardia, sinus disease or other supra-ventricular conduction abnormalities such as sinoatrial or atrioventricular block.
* Taking concomitant medications known to prolong the interval QTc
* Patients at particular risk of ulcer, known ulcer disease or receiving concomitant treatment with non-steroidal anti-inflammatory drugs.
* Patient at risk of urinary retention.
* History of epileptic disease.
* History of neuroleptic malignant syndrome.
* History of asthma or obstructive bronchopulmonary disease.
* Severe hepatic impairment.
* Taking one of the following treatments:

  * CYP3A4 inhibitors, such as ketonazole.
  * 2D6 inhibitors, such as quinidine.
  * CYP3A4 inhibitors, such as itraconazole and erythromycin.
  * CYP2D6 inhibitors, such as fluoxetine.
  * Enzyme inducers such as rifampicin, phenytoin, carbamazepine.
  * Antiarrhythmic class IA agents
  * Antiarrhythmic class III agents
  * other Antipsychotics such as phenothiazine, sertindole, pimozide, ziprasidone.
  * some antiobiotics such as clarithromycine, erythromycine, levofloxacine, moxifloxacine.
* Participation in another interventional study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Difference of change in the MMSE score | 26 weeks
  Difference of change in the MMSE score between baseline and 26 weeks in the 2 ams (donepezil versus non-drug). MMSE is measured at baseline, 6 weeks, 13 weeks, and 26 weeks.

SECONDARY OUTCOMES:
Difference of change in the ADAS-Cog scale | 26 weeks
  Difference of change in the ADAS-Cog scale between baseline and 26 weeks in the 2 ams (donepezil versus non-drug).
  ADAS-Cog scale = Alzheimer's Disease Assessment Scale-Cognitive Subscale, scored from 0 to 70
Difference of change in the CDR scale | 26 weeks
  Difference of change in the CDR scale between baseline and 26 weeks in the 2 ams (donepezil versus non-drug).
  CDR scale = Clinical Dementia Rating, scored from 0 to 3
Difference of change in the ADL scale | 26 weeks
  Difference of change in the ADL scale between baseline and 26 weeks in the 2 ams (donepezil versus non-drug).
  ADL scale = Autonomy scale on daily activities, scored from 0 to 78
Difference of change in the quality of life scale | 26 weeks
  Difference of change in the quality of life scale between baseline and 26 weeks in the 2 ams (donepezil versus non-drug).
Difference of change in the ZARIT scale | 26 weeks
  Difference of change in the ZARIT scale between baseline and 26 weeks in the 2 ams (donepezil versus non-drug).
  ZARIT scale = for assessing caregiver burden, scored from 0 to 88

CONTACTS AND LOCATIONS:
Locations (1):
- Cognitive Neurology Center, Paris, France

IPD SHARING:
Plan to Share IPD: No